CLINICAL TRIAL: NCT02677012
Title: A Randomized, Prospective Comparison of Time Associated With Techniques to Process Autologous Fat Grafts
Brief Title: Autologous Fat Grafting Techniques in Patients Undergoing Reconstructive Surgery
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2015-0006; NCI-2016-00346 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0006 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2016-02-04; First posted 2016-02-09 (Estimated); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Health Status Unknown
MeSH Terms: interventions — Plastic Surgery Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Arm I (RESOLVE TM): Patients undergo AFG reconstructive surgery comprising washing and low velocity spinning using a commercially available system that washes the lipoaspirate with lactated Ringer's solution separates non-fat material from the fat with gentle centrifugal force and suction.
  Interventions: Procedure: Autologous Fat Graft; Procedure: Reconstructive Surgery
- Arm II (Cytori PureGraft TM): Patients undergo AFG reconstructive surgery comprising gravity filtration using a commercially available system in which the lipoaspirate is rinsed with lactated RL and the non-fat material is filtered through mesh.
  Interventions: Procedure: Autologous Fat Graft; Procedure: Reconstructive Surgery
- Arm III (Coleman technique): Patients undergo AFG reconstructive surgery comprising standard centrifugation at 3200 rpm for 3 minutes with the resulting oil and aqueous layers discarded.
  Interventions: Procedure: Autologous Fat Graft; Procedure: Reconstructive Surgery

INTERVENTIONS:
Procedure: Autologous Fat Graft — Undergo AFG using the RESOLVE TM technique
  Other Names: Autologous Fat Cell Transplantation; Autologous Fat Injection; Autologous Fat Transfer
  Groups: Arm I (RESOLVE TM)
Procedure: Autologous Fat Graft — Undergo AFG using the Cytori PureGraft TM technique
  Other Names: Autologous Fat Cell Transplantation; Autologous Fat Injection; Autologous Fat Transfer
  Groups: Arm II (Cytori PureGraft TM)
Procedure: Autologous Fat Graft — Undergo AFG using the Coleman technique
  Other Names: Autologous Fat Cell Transplantation; Autologous Fat Injection; Autologous Fat Transfer
  Groups: Arm III (Coleman technique)
Procedure: Reconstructive Surgery — Undergo reconstructive surgery
  Other Names: Reconstruction

SUMMARY:
This randomized clinical trial studies and compares 3 techniques in performing autologous fat grafting (AFG) in patients undergoing surgery to reshape or rebuild (reconstruct) a part of the body changed by previous surgery and inserted into another part of the body. AFG, also called fat injections or fat transplant, is a procedure in which an individual's own body fat (usually from abdomen or legs) is used during reconstructive surgery. Doctors want to compare 3 techniques for processing the fat tissue collected during surgery and the length of time needed to complete each AFG technique and surgery. Comparing 3 AFG techniques and the time to complete them during surgery may help doctors determine the best technique to perform fat grafting in the future.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Measure and compare the rate of fat processed, defined as the volume of fat processed per unit time associated with the use of three aforementioned adipose tissue processing techniques.

SECONDARY OBJECTIVES:

I. To measure total fat grafting time: time from initiation of fat harvesting to the end of fat injection.

II. To measure volume of fat processed: volume of fat obtained after fat processing.

III. To measure total operation room (OR) time: time from patient entry into the OR (or when the patient barcode is read on entering the OR) to the time at which the patient leaves the OR.

OUTLINE: Patients are randomized to 1 of 3 arms.

ARM I (REVOLVE TM): Patients undergo AFG reconstructive surgery comprising washing and low velocity spinning using a commercially available system that washes the lipoaspirate with lactated Ringer's solution separates non-fat material from the fat with gentle centrifugal force and suction.

ARM II (CYTORI PUREGRAT TM): Patients undergo AFG reconstructive surgery comprising gravity filtration using a commercially available system in which the lipoaspirate is rinsed with lactated Ringer's solution (RL) and the non-fat material is filtered through mesh.

ARM III (COLEMAN TECHNIQUE): Patients undergo AFG reconstructive surgery comprising standard centrifugation at 3200 revolutions per minute (rpm) for 3 minutes with the resulting oil and aqueous layers discarded.

ELIGIBILITY:
Inclusion Criteria:

* Patients with available harvest sites for fat grafting
* Patients with body mass index (BMI) > 20
* Estimated harvested fat volume >= 100 cc
* Patients are willing and able to give consent

Exclusion Criteria:

* Patients with active cancer, including primary cancer, recurrent cancer, or locally or distant metastasis
* Patients who are unable to provide consent
* Patients who are suspected or known to be pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-02-04 (Actual); Primary Completion 2020-07-03 (Actual); Study Completion 2020-07-03 (Actual)

PRIMARY OUTCOMES:
Rate of fat processed defined as the volume of fat harvested per minute | 1 day
  Study data will be collected and managed using the Research Electronic Data Capture. This study will measure and compare the rate of fat processed, defined as the volume of fat processed per unit time associated with the use of three adipose tissue processing techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Summer Hanson, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Hanson SE, Garvey PB, Chang EI, Reece GP, Liu J, Baumann DP, Butler CE. A Randomized Prospective Time and Motion Comparison of Techniques to Process Autologous Fat Grafts. Plast Reconstr Surg. 2021 May 1;147(5):1035-1044. doi: 10.1097/PRS.0000000000007827. PMID 33890883
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org